CLINICAL TRIAL: NCT04919863
Title: A Phase I Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of NTP42:KVA4 in Healthy Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of NTP42:KVA4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ATXA Therapeutics Limited (Industry)
Collaborators: Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ATXA-CT001
Record Dates: First submitted 2021-05-20; First posted 2021-06-09 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NTP42:KVA4 (Experimental)
  Interventions: Drug: NTP42:KVA4
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NTP42:KVA4 — Single ascending dose (SAD) or multiple ascending dose (MAD) of NTP42:KVA4 administered to healthy volunteers as an oral suspension.
  Arms: NTP42:KVA4
Drug: Placebo — Placebo, matched to corresponding doses of NTP42:KVA4 administered to healthy volunteers as an oral solution.
  Arms: Placebo

SUMMARY:
A Phase I clinical trial to assess the safety, tolerability, and pharmacokinetics of NTP42:KVA4 following oral administration in a randomized, double-blind, placebo-controlled trial. The trial will involve of 2 phases, a single ascending dose (SAD) phase and a multiple ascending dose (MAD) phase. The SAD phase will incorporate a food effect arm.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI) in the range 18.0-30.0.
* Ability & willingness to provide written consent.

Exclusion Criteria:

* Clinically relevant abnormal medical history, physical findings, laboratory values at pre-trial screening.
* History of bleeding disorders, coagulation variables or abnormal blood cell count.
* History of chronic illness.
* Impaired endocrine, thyroid, hepatic, renal or respiratory function, diabetes mellitus, coronary heart disease or history of any psychotic mental illness.
* History of adverse reaction or allergy to any drug.
* Use of aspirin, other non-steroidal anti-inflammatory drugs (NSAIDs), or any other medicine that affects platelet function or coagulation, or any prescription medicine, during the 28 days before the first dose of trial medication.
* History of drug or alcohol abuse
* Smoker or use of nicotine-containing products
* Blood pressure or heart rate at screening outside normal ranges.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of single and repeated doses of NTP42:KVA4 in healthy volunteers. | Up to 48-hour post-dose.
  Adverse events (AEs)
Evaluation of the pharmacokinetics of single and repeated doses of NTP42:KVA4 in healthy volunteers. | Predose, 0.16, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 18, 24, 36 & 48 hours post-dosing.
  Pharmacokinetic parameter: Area under the Curve (AUC)
Evaluation of the effect of food on the pharmacokinetics of NTP42:KVA4 in healthy volunteers. | Predose, 0.16, 0.5, 0.75, 1, 2, 4, 6, 8, 12, 18, 24, 36 & 48 hours post-dosing.
  Pharmacokinetic parameter: Area under the Curve (AUC)

SECONDARY OUTCOMES:
Evaluation of the pharmacodynamics effects of NTP42:KVA4 in healthy volunteers. | Predose, 0.75, 2, 4, 8, 12 & 24 hours post-dosing
  TXA2-induced platelet aggregometry

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Boyce, MD, Principal Investigator — Hammersmith Medicines Reserach
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

REFERENCES:
- [Derived] Reid HM, Maginn M, Perkins CM, Mulvaney EP, Boyce M, Yamamoto T, Kinsella BT. Evaluation of NTP42, a novel thromboxane receptor antagonist, in a first-in-human phase I clinical trial. Front Pharmacol. 2023 Dec 21;14:1296188. doi: 10.3389/fphar.2023.1296188. eCollection 2023. PMID 38178863